CLINICAL TRIAL: NCT01356082
Title: Accuracy of the CNAP™ Monitor in Providing Beat-to-beat Non-invasive Blood Pressure Readings
Brief Title: CNAP™ Monitor Study
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB11-00170
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Cardiac Surgery; Spinal Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arterial blood pressure line: Patients receiving an arterial blood pressure line
  Interventions: Device: CNAP

INTERVENTIONS:
Device: CNAP — Non-invasive blood pressure monitor

SUMMARY:
A newly developed monitor for continuous non-invasive blood pressure monitoring (CNAP™ Monitor 500; CNSystems Medizintechnik AG, Graz, Austria) provides beat-to-beat BP readings and is non-invasive. To make sure that anaesthesiologist can rely on and make clinical decisions based on values provided by the CNAP™ monitor, to demonstrate its reliability we will test it during the perioperative care of children.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will already be having an indwelling arterial cannula placed for their surgical procedure.

Exclusion Criteria:

* Patients with history of a peripheral neurologic or neuropathic disorder.
* Patients in whom an invasive arterial cannula cannot be placed.
* Patients with vascular implants at the sites of non-invasive blood pressure measurement (fingers and upper arm of the examined arm).
* Edematous patients.
* Patients who are less than 20 kg.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Surgery patients at Nationwide Children's Hospital receiving an arterial line.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 1 Day (day of surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States